CLINICAL TRIAL: NCT01826526
Title: Taurolidine 2% Catheter Locking to Prevent Catheter-related Bloodstream Infections in Patients on Home Parenteral Nutrition With a High Infection Risk and Those With a New Central Venous Access Device
Brief Title: Clinical Trial With Catheter Locking TauroSept® (Taurolidine 2%) or Saline Solution 0,9%
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geert Wanten (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Geert Wanten, MD, PhD, MSc, Radboud University Medical Center
Organization: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TCL-0112
Record Dates: First submitted 2013-03-05; First posted 2013-04-08 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Catheter Related Blood Stream Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TauroSept® (Active Comparator): 5 ml of TauroSept® will be instilled into the catheter (CVAD) each time after total parenteral nutrition (TPN) has been completed. The frequency of administration depends on the schedule of HPN. It varies between twice per week and once daily.
  The duration of TauroSept® administration in this trial will be 12 months.
  Interventions: Device: TauroSept®
- Saline solution 0.9% (Placebo Comparator): 5 ml of saline will be instilled into the catheter (CVAD) each time after total parenteral nutrition (TPN) has been completed. The frequency of administration depends on the schedule of HPN. It varies between twice per week and once daily.
  The duration of saline administration in this trial will be 12 months.
  Interventions: Device: TauroSept®

INTERVENTIONS:
Device: TauroSept® — 5 ml of TauroSept® will be instilled into the catheter (CVAD) each time after total parenteral nutrition (TPN) has been completed. The frequency of administration depends on the schedule of HPN. It varies between twice per week and once daily.
  The duration of TauroSept® administration in this trial will be 12 months.
  Other Names: Taurolidine 2%

SUMMARY:
The purpose of this study is to determine if TauroSept® taurolidine 2% is more efficient than saline solution 0.9% as a catheter lock solution in preventing catheter related blood stream infections in patients with home parenteral nutrition.

DETAILED DESCRIPTION:
Home Parenteral Nutrition has become a mainstay in the support of patients with chronic intestinal failure. It requires the presence of a central venous catheter to assure adequate venous access. Catheter Related BloodStream Infections (CRBSIs) are frequent. Most CRBSIs originate from contamination of the catheter hub and subsequent growth of microorganisms embedded within the biofilm that rapidly develops on the inner catheter surface. The best preventive measure against the development of CRBSIs is observation of strict hygiene guidelines when inserting and manipulating a central venous catheter and in addition to this the instillation of antimicrobial solutions like TauroSept® or saline solution 0.9% into the catheter lumen (antimicrobial lock). This measure is currently widely used in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Benign underlying disease leading to long-term intestinal failure who will receive HPN and/or fluids (saline and/or glucose) at least 2 times /week over a subcutaneously tunnelled single-lumen Central Venous Catheter (CVC) (Hickman/Broviac or subcutaneous port) for at least one year

  1. Patient receives a new single lumen central vascular access device for HPN (new patient starting HPN or patient already on HPN) allocation to Group I = new catheter group] or
  2. Patient is already on HPN for ≥1 year prior to trial inclusion and has a CRBSI rate (bacterial and/or yeast infections) of >0.3/year and a catheter that has been in place for ≥6 months (allocation to Group II = high risk group). (Previous salvage of this catheter by line-lock antibiotics or other therapeutic interventions is not an exclusion criterion as long as this has been performed at least two months before enrolment in the trial)
* Estimated life expectancy ≥1 year
* Male or female patient aged 18 - 80 years
* Patient is fully able to understand the nature of the proposed intervention and gives written informed consent before entering the trial.

Exclusion Criteria:

* cannot be expected to comply with the trial plan (substance abuse, mental condition)
* has significant cardiovascular disease such as unstable angina, acute myocardial infarction or recent cerebral vascular accident (within 6 weeks); a cardiac rhythm which in the investigators judgment may result in significant hemodynamic effects
* has a known hypersensitivity/allergy to taurolidine 2% or saline solution 0.9% and/or their excipients.
* is pregnant, lactating, or nursing.
* has a current bloodstream infection
* has any clinically significant abnormalities in blood coagulation requiring intervention
* has received thrombolytic therapy in the 6 weeks prior to insertion (aspirin 80-325 mg daily is acceptable).
* has received an investigational drug within 30 days of trial entry
* has an antibiotic coated, silver impregnated or antimicrobial cuff catheter
* has received a Taurolidine lock previously
* has compromised skin integrity, including any infection at the insertion site
* has received parenteral or oral antibiotic therapy <2months prior trial inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-06; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Mean number of catheter related blood stream infections CRBSI/1'000 catheter days in each group | 12 months

SECONDARY OUTCOMES:
Median time to a catheter related blood stream infection CRBSI per patient per group | 12 months

CONTACTS AND LOCATIONS:
Locations (7):
- University Hospital Copenhagen Rigshospitalet, Copenhagen, Denmark
- University Clinic Münster, Münster, Germany
- Rabin Medical Center, Petah Tikva, Israel
- University of Bologna Center for Chronic Intestinal Failure Department of Gastroenterology and Internal Medicine, Bologna, Italy
- Department of Gastroenterology and Hepatology clinical ward, Nijmegen, Netherlands
- United Kingdom (2):
  - St Mark's Hospital, Harrow, Middlesex
  - University College Hospital, London

REFERENCES:
- [Result] Bisseling TM, Willems MC, Versleijen MW, Hendriks JC, Vissers RK, Wanten GJ. Taurolidine lock is highly effective in preventing catheter-related bloodstream infections in patients on home parenteral nutrition: a heparin-controlled prospective trial. Clin Nutr. 2010 Aug;29(4):464-8. doi: 10.1016/j.clnu.2009.12.005. Epub 2010 Jan 12. PMID 20061070
- [Derived] Wouters Y, Theilla M, Singer P, Tribler S, Jeppesen PB, Pironi L, Vinter-Jensen L, Rasmussen HH, Rahman F, Wanten GJA. Randomised clinical trial: 2% taurolidine versus 0.9% saline locking in patients on home parenteral nutrition. Aliment Pharmacol Ther. 2018 Aug;48(4):410-422. doi: 10.1111/apt.14904. Epub 2018 Jul 5. PMID 29978597
- [Derived] Tribler S, Brandt CF, Fuglsang KA, Staun M, Broebech P, Moser CE, Scheike T, Jeppesen PB. Catheter-related bloodstream infections in patients with intestinal failure receiving home parenteral support: risks related to a catheter-salvage strategy. Am J Clin Nutr. 2018 May 1;107(5):743-753. doi: 10.1093/ajcn/nqy010. PMID 29722835